CLINICAL TRIAL: NCT04730921
Title: Impact of Left Bundle Branch Area Pacing vs. Right Ventricular Pacing in Atrioventricular Block (LEAP-Block): A Randomized Controlled Trial
Brief Title: Impact of Left Bundle Branch Area Pacing vs. Right Ventricular Pacing in Atrioventricular Block (LEAP-Block)
Acronym: LEAP-Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Wai Hospital, Beijing, China (Other)
Collaborators: Beijing Anzhen Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); The Second Hospital of Hebei Medical University (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Tianjin Medical University General Hospital (Other); TEDA International Cardiovascular Hospital (Other); Peking Union Medical College Hospital (Other); Chinese Society of Cardiology (Other); Affiliated Hospital of Qinghai University (Other); Shanxi Cardiovascular Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); Peking University First Hospital (Other); Beijing Friendship Hospital (Other); Wuxi People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaohan Fan, Professor, MD, PhD, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-1379
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-07

CONDITIONS: Atrioventricular Block; Left Bundle Branch Area Pacing; Right Ventricular Pacing; Heart Failure
Keywords: Atrioventricular Block; Left bundle branch area pacing; Right ventricular pacing
MeSH Terms: conditions — Atrioventricular Block; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- LBBAP group (Experimental): AV block patients randomized to left bundle branch area pacing
  Interventions: Device: Left bundle branch area pacing
- RVP group (Active Comparator): AV block patients randomized to right ventricular pacing group
  Interventions: Device: Right ventricular pacing

INTERVENTIONS:
Device: Left bundle branch area pacing — Left bundle branch area pacing(LBBAP) is a novel physiological pacing form for ventricular pacing. In patients received LBBAP, the pacing lead will be placed at left bundle branch area to achieve narrow paced QRS duration.
  Arms: LBBAP group
Device: Right ventricular pacing — Right ventricular pacing is the traditional pacing modality for ventricular pacing. The pacing lead was placed in the apex or septum of right ventricle.
  Arms: RVP group

SUMMARY:
This is a multicenter, randomized controlled study. The aim of this study is to compare the impact of LBBAP on left ventricular function as compared with traditional right ventricular pacing in patients with atrioventricular block.

DETAILED DESCRIPTION:
LEAP-BLOCK is a prospective, multi-center, randomized controlled trial that is designed to determine whether left bundle branch area pacing (LBBAP) may reduce the risk of RV ventricular pacing induced cardiac dysfunction as compared with traditional RV pacing (RVP) in patients with atrioventricular (AV) block and normal LV function (LVEF≥50%) who require high percent of ventricular pacing. The primary aim of this trial is to compare the time to first event (composite of all-cause mortality and newly heart failure hospitalization and device upgrade due to heart failure) between LBBAP and RVP group in patients with AV block. Patients with AV block and normal LV function who require high burden of ventricular pacing (expected >40%) will be randomized to LBBAP or RVP group for therapy. Patients will be followed at least every 3 months for clinical status and every 6 months for echocardiographic evaluation until the study closure.

ELIGIBILITY:
Inclusion Criteria:

* a. Adult patients aged 18-90;
* b. AV block patients with ventricular pacing indications and the expected rate of ventricular pacing(VP)> 40%, including (a)Third-degree AV block; (b) Second degree AV block (type II); (c) intermittent advanced AV block with expected VP>40%; (d)Symptomatic first degree AV block and PR interval on ECG ≥ 250ms;
* c. The subject is able to receive a pectoral implant;
* d. The subject is willing and able to comply with the protocol;
* e. The subject is expected to remain available for follow-up visits at the study centers.
* f. Subject or authorized legal guardian or representative has signed and dated the study Subject Informed Consent

Exclusion Criteria:

* a. Baseline echocardiographic assessment of patients with impaired LV function (LVEF<50%);
* b. Having difficulties in follow-up: Those who cannot accept 2-year follow-up on time due to physical condition or other reasons;
* c. Patients with persistent atrial fibrillation;
* d. Pacemaker replacement without new implanted ventricular electrodes;
* e. Patients with implantable cardioverter-defibrillator (ICD) indications;
* f. Surgery is required within 1 year due to severe structural heart disease;
* g. Patients with tricuspid mechanical valve replacement, or congenital heart disease (including transposition of the great arteries, or permanent left superior vena cava, etc), or AV block resulting from: (a) Hypertrophic cardiomyopathy(HCM)vpost (modified) Morrow surgery, (b) ventricular septal defect repair; and those who are unlikely to achieve successful LBBAP procedure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the time to a first event of composite outcomes, including all-cause death, hospitalization for heart failure, and an upgrade to cardiac resynchronization therapy due to pacing induced heart failure. | Within two years after device implantation
  All-cause death: including cardiovascular and non-cardiovascular deaths. Hospitalization for heart failure: an unplanned outpatient or emergency department visit or inpatient hospitalization in which the patient presented with signs and symptoms consistent with heart failure and required medication therapy.
  Upgrade to cardiac resynchronization therapy (CRT): Upgrade from dual-chamber pacemaker to CRT-Pacemaker/CRT-Defibrillator due to impaired LV function (LVEF decrease to 40% or less).

SECONDARY OUTCOMES:
Rate of the composite outcomes of all-cause death and/or hospitalization for heart failure | Within 2 years after device implantation
  All-cause death: including cardiovascular and non-cardiovascular deaths. Hospitalization for heart failure: an unplanned outpatient or emergency department visit or inpatient hospitalization in which the patient presented with signs and symptoms consistent with heart failure and required medication therapy.
Rate of the composite outcomes of hospitalization for heart failure and/or an upgrade to cardiac resynchronization therapy due to pacing induced heart failure. | Within 2 years after device implantation
  Hospitalization for heart failure: an unplanned outpatient or emergency department visit or inpatient hospitalization in which the patient presented with signs and symptoms consistent with heart failure and required medication therapy.
  Upgrade to cardiac resynchronization therapy: Upgrade from dual chamber pacemaker to CRT-P/CRT-D due to impaired LV function (LVEF decrease to 40% or less).
Rate of the composite outcomes of LVEF <50%, and/or an increase in LVESV ≥15% during follow-up as compared with the value at randomization | Within 2 years after device implantation
  Echocardiography will be assessed every 6 month during follow-up to determine whether the LVEF is less than 50% and/or the LVESV is increased by 15% or more.
The value of LVEF and LVESV assessed by echocardiography at 1-year and 2-year follow-up | 24 months
  Echocardiography will be assessed at 1-year, and 2-year follow-up and the absolute value of LVEF and LVESV will be compared between two groups.
The time to a first event of LVEF <50% and decrease in LVEF by ≥ 10% during 2 years follow-up as compared with the value at randomization. | 24 months
  Echocardiography will be assessed every 6 month during follow-up to determine whether the LVEF is less than 50% and decreased by 15% or more as compared with the value at randomization.
The immediate success rate of the LBBAP procedure | 1 weeks
  Successful LBBAP procedure is identified according to ECG and intracardiac electrogram (IEGM) during the procedure. All LBBAP procedures will be categorized as selective left bundle branch pacing (S-LBBP), non-selective left bundle branch pacing(NS-LBBP), or left ventricular septal pacing (LVSP).
The rate of procedure and Device related complications | 24 months
  Procedure complications include pneumothorax, hemothorax, and air embolism. Device related complications include lead and pocket complications.
Changes in Pacing parameters and ECG characteristics. | 24 months
  Pacing parameters include pacing thresholds (ventricle), Sense ampitude (ventricle), Impedance (ventricle). ECG characteristics include paced QRS duration and QRS morphology, etc.
The occurrence of LV dyssynchrony | 24 months
  The occurrence of LV dyssynchrony will be evaluated by echocardiography during 2-year follow-up.
Atrial high-rate episodes recorded by the pacemaker | 24 months
  Atrial high-rate episodes recorded in the pacemaker will be followed during two years of follow-up
The long-term success rate of LBBAP | 24 months
  In LBBAP group, the successful LBBAP will be identified according ECG features at 2-years follow-up

OTHER OUTCOMES:
Pre-existing heart disease based primary outcome | Within 2 years after device implantation
  All-cause death and/or hospitalization for heart failure comparison based on pre-exsiting heart disease (e.g. coronary heart disease, atrial fibirllation, valvular heart disease, and dilated cardiomyopathy.
Baseline QRSd based primary outcome | Within 2 years after device implantation
  All-cause death and/or hospitalization for heart failure comparison based on baseline QRSd (>120ms vs. ≤120ms)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohan Fan, PhD., Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (8):
- China (8):
  - Beijing Anzhen hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Teda International Cardiovascular Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu CM, Chan JY, Zhang Q, Omar R, Yip GW, Hussin A, Fang F, Lam KH, Chan HC, Fung JW. Biventricular pacing in patients with bradycardia and normal ejection fraction. N Engl J Med. 2009 Nov 26;361(22):2123-34. doi: 10.1056/NEJMoa0907555. Epub 2009 Nov 15. PMID 19915220
- [Background] Vijayaraman P, Naperkowski A, Subzposh FA, Abdelrahman M, Sharma PS, Oren JW, Dandamudi G, Ellenbogen KA. Permanent His-bundle pacing: Long-term lead performance and clinical outcomes. Heart Rhythm. 2018 May;15(5):696-702. doi: 10.1016/j.hrthm.2017.12.022. Epub 2017 Dec 20. PMID 29274474
- [Background] Cho SW, Gwag HB, Hwang JK, Chun KJ, Park KM, On YK, Kim JS, Park SJ. Clinical features, predictors, and long-term prognosis of pacing-induced cardiomyopathy. Eur J Heart Fail. 2019 May;21(5):643-651. doi: 10.1002/ejhf.1427. Epub 2019 Feb 8. PMID 30734436
- [Background] Tayal B, Fruelund P, Sogaard P, Riahi S, Polcwiartek C, Atwater BD, Gislason G, Risum N, Torp-Pedersen C, Kober L, Kragholm KH. Incidence of heart failure after pacemaker implantation: a nationwide Danish Registry-based follow-up study. Eur Heart J. 2019 Nov 21;40(44):3641-3648. doi: 10.1093/eurheartj/ehz584. PMID 31504437
- [Background] Huang W, Su L, Wu S, Xu L, Xiao F, Zhou X, Mao G, Vijayaraman P, Ellenbogen KA. Long-term outcomes of His bundle pacing in patients with heart failure with left bundle branch block. Heart. 2019 Jan;105(2):137-143. doi: 10.1136/heartjnl-2018-313415. Epub 2018 Aug 9. PMID 30093543
- [Background] Abdelrahman M, Subzposh FA, Beer D, Durr B, Naperkowski A, Sun H, Oren JW, Dandamudi G, Vijayaraman P. Clinical Outcomes of His Bundle Pacing Compared to Right Ventricular Pacing. J Am Coll Cardiol. 2018 May 22;71(20):2319-2330. doi: 10.1016/j.jacc.2018.02.048. Epub 2018 Mar 10. PMID 29535066
- [Background] Vijayaraman P, Dandamudi G. Anatomical approach to permanent His bundle pacing: Optimizing His bundle capture. J Electrocardiol. 2016 Sep-Oct;49(5):649-57. doi: 10.1016/j.jelectrocard.2016.07.003. Epub 2016 Jul 11. PMID 27457727
- [Background] Li X, Li H, Ma W, Ning X, Liang E, Pang K, Yao Y, Hua W, Zhang S, Fan X. Permanent left bundle branch area pacing for atrioventricular block: Feasibility, safety, and acute effect. Heart Rhythm. 2019 Dec;16(12):1766-1773. doi: 10.1016/j.hrthm.2019.04.043. Epub 2019 Apr 29. PMID 31048065
- [Background] Li X, Qiu C, Xie R, Ma W, Wang Z, Li H, Wang H, Hua W, Zhang S, Yao Y, Fan X. Left bundle branch area pacing delivery of cardiac resynchronization therapy and comparison with biventricular pacing. ESC Heart Fail. 2020 Aug;7(4):1711-1722. doi: 10.1002/ehf2.12731. Epub 2020 May 13. PMID 32400967
- [Background] Sharma PS, Dandamudi G, Naperkowski A, Oren JW, Storm RH, Ellenbogen KA, Vijayaraman P. Permanent His-bundle pacing is feasible, safe, and superior to right ventricular pacing in routine clinical practice. Heart Rhythm. 2015 Feb;12(2):305-12. doi: 10.1016/j.hrthm.2014.10.021. Epub 2014 Oct 22. PMID 25446158